CLINICAL TRIAL: NCT06097936
Title: New Prognostic and Predictive Biomarkers for HPV-associated Oropharyngeal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: University of California, San Diego (Other); Lega Italiana per la Lotta contro i Tumori (Other)
Responsible Party: Sponsor
Other Study IDs: RS1443/20(2442)
Record Dates: First submitted 2023-03-28; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-06

CONDITIONS: PREDICTIVE BIOMARKERS; Evaluation of HPV-specific E5 Transcript Expression in a Cohort of Patients With HPV-associated OPC; HPV 16 Positive Oropharyngeal Tumors (OPC)
Keywords: HPV 16; oropharyngeal tumors (OPC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HPV Patients
  Interventions: Diagnostic Test: HPV-ASSOCIATED OROPHARYNGEAL CANCER

INTERVENTIONS:
Diagnostic Test: HPV-ASSOCIATED OROPHARYNGEAL CANCER — The study involves the coexistence of a retrospective part, in which a group of patients with HPV-associated OPC for whom follow-up data of at least 2 years after diagnosis are available, designed in order to evaluate the expression of HPV16-specific E5 transcript as well as that of pEGFR and HLA, and a multicenter prospective part, involving the enrollment of a control group, enrolled at the ENT outpatient clinic of the IRE and the outpatient clinics of the relevant LILT provincial committees, to better elucidate the role of HPV16-E5 in identifying potentially transforming infections due to the presence of HPV.

SUMMARY:
The study involves the coexistence of a retrospective part, in which a group of patients with HPV-associated OPC for whom follow-up data of at least 2 years after diagnosis are available, designed in order to evaluate the expression of HPV16-specific E5 transcript as well as that of pEGFR and HLA, and a multicenter prospective part, involving the enrollment of a control group, enrolled at the ENT outpatient clinic of the IRE and the outpatient clinics of the relevant LILT provincial committees, to better elucidate the role of HPV16-E5 in identifying potentially transforming infections due to the presence of HPV.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* age > 18 years
* current and/or former smokers
* reporting at least 5 (Souza 2017) lifetime oral sex partners
* Written informed consent

Exclusion Criteria:

* Oral pathology
* inability to understand and sign an informed consent form

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group will be enlisted from among the subjects referred to the IRE outpatient clinic and/or the outpatient clinics of the LILT Provincial Committees collaborating with the Project to undergo a screening/checkup visit.
  Samples will be collected in a mouthwash (i.e., Listerine) and stored in suitable solution to preserve nucleic acids (i.e., PreservCyt Transport Medium) and sent by courier from the peripheral centers to the IFOs where they will be appropriately analyzed.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Presence of specific mRNA for the E5 oncoprotein in HPV-associated OPC samples | Sample collection period: 6 months Total duration of the study: 12 months
  The expected results concern the identification of OPC subgroups correlated with the expression of HPV16 E5.RNA will be extracted from FFPE with a commercial RNeasy kit (QIAGEN) and reverse transcribed into cDNA.
  The synthesized cDNA will be subjected to real-time PCR with specific primers, already designed by the Beacon Design software (BioRad) to include the splicing site (880-3358) of the specific E5 transcript.
  The relative amount of genes will be determined by the ΔΔCt method normalized to housekeeping genes.

SECONDARY OUTCOMES:
Presence of specific mRNA for the E5 oncoprotein in HPV-associated OPC samples | Sample collection period: 6 months Total duration of the study: 12 months
  the primary outcome is necessary for a subsequent larger study in which the expression of E5 will be evaluated together with that of EGFR and HLA and associated with prognosis and different responses to therapy

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided